CLINICAL TRIAL: NCT01509092
Title: Traumatic Macular Hole: Six-months Observation Versus Early Surgical Intervention, A Multicenter Clinical Trial
Brief Title: Comparative Study Between Early Vitrectomy and Observation for Spontaneous Closure of Traumatic Macular Hole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Zhi-zhong Ma, Professor, Peking University Third Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PekingUTH-TMH-2011
Record Dates: First submitted 2011-12-28; First posted 2012-01-12 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2012-01

CONDITIONS: Trauma; Macular Hole
Keywords: traumatic macular hole; vitrectomy; observation
MeSH Terms: conditions — Wounds and Injuries; Retinal Perforations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- obervation (No Intervention): patients in this arm received 6-months observation alone after injury
- Surgical intervention (Active Comparator): patients in this arm received vitrectomy surgery as soon as possible after injury
  Interventions: Procedure: vitrectomy surgery

INTERVENTIONS:
Procedure: vitrectomy surgery — "pars plana vitrectomy +internal limiting membrane peeling" done immediately after the identification of the macular hole
  Arms: Surgical intervention

SUMMARY:
The purpose of this study is to compare the anatomical and visual recovery of eyes with traumatic macular hole (TMH) following either early vitrectomy or 6-month observation.

DETAILED DESCRIPTION:
Patients who received vitrectomy immediately after the injury were compared with patients who were observed for six months for spontaneously closure.The closure rate, foveal microstructure, and final visual acuity were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* closed globe injury
* identification of full-thickness macular hole by optical coherence tomography within one month after trauma

Exclusion Criteria:

* open globe injury
* coexistence of idiopathic macular hole
* severe opaque in the visual axis caused by the injury(eg. severe cataract, severe vitreous hemorrhage)
* combined injuries requiring immediate surgical intervention (eg. lens dislocation, retinal detachment, cyclodialysis)
* coexistence of high myopia
* coexistence of choroidal rupture or subretinal hemorrhage within the diameter of 400μm from the center of the foveola
* coexistence of severe optic nerve injury (no light perception, positive afferent pupillary defect)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
macular hole closure rate | 6 month after injury

SECONDARY OUTCOMES:
central foveal thickness | 6 month after hole closure
length of inner-segment outer-segment junction defect | 6 month after hole closure
final visual acuity | 6 month after hole closure

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Zhong Ma, M.D., Principal Investigator — Peking University Third Hospital
Locations (8):
- China (8):
  - Eye Hospital of Hebei Province, Xingtai, Hebei
  - Weifang Eye Hospital, Weifang, Shandong
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Wenzhou Medical College, Wenzhou, Zhejiang
  - China - Japan Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Southwest Eye hospital of Third Military Medical University, Chongqing
  - Shanghai Ninth People's Hospital Affiliated Shanghai JiaoTong University school of Medicine, Shanghai